CLINICAL TRIAL: NCT04426864
Title: Efficacy of Different Types of Exercises on Pain, Quality of Life, Depression, and Body Composition in Women With Fibromyalgia Syndrome.
Brief Title: Efficacy of Different Types of Exercises in Women With Fibromyalgia Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Füsun Ardıç, Director, Head of Physical Medicine and Rehabilitation, Principal Investigator, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018TIPF044
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia; Aerobic exercise; Resistance exercise; Stretching exercise
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Participants are assigned to three groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Aerobic Plus Stretching Exercises Group (Active Comparator): The participants were instructed to perform the walking exercise at their target HR on a treadmill and stretching exercises before and after the exercise program in the Sports Rehabilitation Unit of Pamukkale University.
  Interventions: Other: Supervised Aerobic Plus Stretching Exercises
- Supervised Resistance Plus Stretching Exercises Group (Experimental): The participants were instructed to perform resistance exercises using weight machines and stretching exercises before and after the exercise program in the Sports Rehabilitation Unit of Pamukkale University.
  Interventions: Other: Supervised Resistance Plus Stretching Exercises Group
- Home-based Stretching Exercises Group (Experimental): The participants were instructed to perform the stretching exercises at home.
  Interventions: Other: Home-based Stretching Exercises Group

INTERVENTIONS:
Other: Supervised Aerobic Plus Stretching Exercises — An exercise prescription was developed for each woman based on the data acquired from the baseline treadmill exercise test. Target HR corresponding to values of 50-70 % ergospirometric VO2max (moderate-intensity) was determined by the submaximal treadmill test. The participants were instructed to perform their exercises at 50 % of VO2max for six weeks. At seventh their exercise intensity was increased to target HR corresponding to 70 % of VO2max. HR was monitored by a Polar HR monitor (Polar Beat, Port Washington, NY). Stretching exercises were performed at the beginning and end of each exercise session. Each muscle group exercise was performed 3-4 times and each repeat was 30 seconds long. The muscle groups which were involved in stretching exercises were upper trapezius, rhomboid, hip flexor, hamstring, pectoral, piriformis, quadriceps, gastrocnemius, soleus, levator scapulae, hip adductor and tensor fasciae late muscles. The exercise program was applied 3 days a week for 12 weeks.
  Arms: Supervised Aerobic Plus Stretching Exercises Group
Other: Supervised Resistance Plus Stretching Exercises Group — According to the data obtained from 1-RM tests, an exercise prescription was developed for each woman. The participants were instructed to perform their exercises with 50% of 1-RM for six weeks. In the 7. week, weights were increased to 70-80% of 1-RM. The number of sets increased progressively (10 repetitions per set; 1 set in the first two weeks; 2 sets in the 3rd and 4th week; 3 sets in the 5th and 6th week). The muscle groups which were involved in resistance exercises were bilateral biceps, deltoid, trapezius, pectorals, serratus anterior, latissimus dorsi, levator scapulae, rhomboid, gluteal, quadriceps, hip adductor and abductor, hamstring, gastrocnemius and abdominal muscles. Stretching exercises were performed at the beginning and end of each exercise session. Each muscle group exercise was performed 3-4 times and each repeat was 30 seconds long. Stretching exercises were given for the muscle groups they worked on. The exercise program was applied 3 days a week for 12 weeks.
  Arms: Supervised Resistance Plus Stretching Exercises Group
Other: Home-based Stretching Exercises Group — Each exercise was described to the patient by visually. For each muscle group exercise was performed for 3-4 times and each repeat was 30 seconds long. The muscle groups which were involved in stretching exercises were upper trapezius, rhomboid, hip flexor, hamstring, pectoral, piriformis, quadriceps, gastrocnemius, soleus, levator scapulae, hip adductor and tensor fasciae late muscles. Exercise program was applied 3 days in a week during 12 weeks. Each participant was called every 2 weeks to maintain compliance.
  Arms: Home-based Stretching Exercises Group

SUMMARY:
Objective: To demonstrate the most effective exercise intervention for women with fibromyalgia syndrome on the pain, quality of life, depression, and body composition through a comparative study of three types of exercise intervention: supervised aerobic plus stretching, supervised resistance plus stretching, and home-based stretching.

DETAILED DESCRIPTION:
Objective: To demonstrate the most effective exercise intervention for women with fibromyalgia syndrome on the pain, quality of life, depression, and body composition through a comparative study of three types of exercise intervention.

Methods: Eighty-four patients women with fibromyalgia syndrome were assigned to three groups: supervised aerobic plus stretching exercises group (group I, n:28), supervised resistance plus stretching exercises group (group II, n:28) and home-based stretching exercises group (group III, n:28). The target heart rate (HR) corresponding to values of 50-70 % ergospirometric VO2max were determined by the submaximal treadmill test. Group I was instructed walking at their target HR on a treadmill. Exercise intensity in group II was determined by one-repetition maximum (1RM) measurements. Group III was instructed to exercise at home. All participants were instructed to perform stretching exercises. Before and after a 12-week exercise program, participants were evaluated by weight, Body Mass Index (BMI), total body fat and muscle percentage, Visual Analog Scale (VAS), Fibromyalgia Impact Questionnaire (FIQ), Short Form-36 (SF-36) and Beck Depression Inventory (BDI).

Study Type: Interventional (Clinical Trial)

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants who meet the criteria for inclusion were women with Fibromyalgia Syndrome diagnosis according to ACR 2016 Fibromyalgia Diagnostic Criteria and were 18-65 years old.
* Participants were well communicative, motivated, and willing to participate in the study.

Exclusion Criteria:

• The exclusion criteria were the presence of uncontrolled hypertension, history of myocardial infarction or coronary artery disease, unstable angina pectoris, class 3-4 heart failure (New York Heart Association), musculoskeletal or systemic diseases contradicting the exercise, a neurological or psychiatric disease affecting cooperation and cognitive function, presence of active inflammation and immunosuppression.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on the self-representation of gender identity.
Enrollment: 84 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in analogue scale (VAS) score at week 12 | Week 12
  Pain intensity was measured with VAS for pain (0-10 cm; 0: no pain, 10: severe pain).
Change from baseline in Fibromyalgia Impact Questionnaire (FIQ) score at week 12 | Week 12
  The Fibromyalgia Impact Questionnaire was designed to measure the health status of patients with fibromyalgia. Total score range from 0 to 100, with higher scores indicating higher levels of symptoms and severity.
Change from baseline Beck Depression Inventory (BDI) score (0-63) at week 12 | Week 12
  This is a 21-item questionnaire that investigates the symptoms of depression. Total score range from 0 to 63, higher scores indicate higher levels of depression.
Change from baseline in Short Form 36 (SF-36) score at week 12. | Week 12
  Short- form health survey 36 contains 36 items which are used to evaluate the quality of life of patients. It measures eight different domains that address physical functioning, physical role limitation, body pain, general health, vitality, social functioning, emotional role limitation and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life).
Change from baseline in weight (kilograms) at week 12. | Week 12
  Weight was measured with body composition analyzer (Tanita MC580).
Change from baseline in body mass index (BMI) at week 12 | Week 12
  Height was measured with stadiometer and BMI was calculated with body composition analyzer (Tanita MC580).
Change from baseline in total body fat percentage at week 12 | Week 12
  Total body fat percentage was measured with body composition analyzer (Tanita MC580).
Change from baseline in in total body muscle percentage at week 12. | Week 12
  Total body muscle percentage was measured with body composition analyzer (Tanita MC580).
Change from baseline in blood lactate concentration at rest (mmol/L) at week 12 | Week 12
  Finger-stick capillary whole blood was collected at rest. Blood lactate concentration was performed using a lactate analyzer (Lactate Scout Plus)

CONTACTS AND LOCATIONS:
Overall Officials: Fusun ARDIC, Prof.M.D., Study Director — Pamukkale University
Locations (1):
- Pamukkale University Faculty of Medicine, Denizli, Turkey (Türkiye)